CLINICAL TRIAL: NCT03250572
Title: Serum Ferritin as a Non-invasive Marker in Prediction of Hepatic Fibrosis Among Non-alcoholic Fatty Liver Disease Patients
Brief Title: Serum Ferritin as a Non-invasive Marker in Prediction of Hepatic Fibrosis Among NAFLD Patients
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shereen Abou Bakr Saleh, Asisstant Professor, Ain Shams University
Other Study IDs: 9875
Record Dates: First submitted 2017-08-08; First posted 2017-08-15 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- control group
  Interventions: Diagnostic Test: serum ferritin
- NAFLD patients without hepatic fibrosis
  Interventions: Diagnostic Test: serum ferritin
- NAFLD patients with hepatic fibrosis
  Interventions: Diagnostic Test: serum ferritin

INTERVENTIONS:
Diagnostic Test: serum ferritin — serum samples and ferritin ELISA test

SUMMARY:
This study was designed to assess the relation between serum ferritin and hepatic fibrosis in patients with NAFLD. It included 83 patients with NAFLD with or without hepatic fibrosis, in addition to 30 healthy subjects included as controls. Measurement of serum ferritin and its correlation with steatosis and fibrosis was done.

DETAILED DESCRIPTION:
Background: many studies have found a relationship between hepatic iron, serum ferritin and NAFLD or its progress. Aim of the work: is to assess the value of serum ferritin as a non-invasive marker in prediction of hepatic fibrosis in NAFLD. Methods: This study included 113 subjects who were classified into 3 groups. Group I: included 30 healthy subjects as control with no evidence of NAFLD by liver biopsy. Group II: included 31 NAFLD patients without fibrosis proved by liver biopsy. Group III: included 52 patients with hepatic fibrosis on top of NAFLD proved by liver biopsy. Serum ferritin was determined using Ferritin ELISA kit. FIB4 was calculated and liver biopsy was done for all patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with NAFLD with or without hepatic fibrosis

Exclusion Criteria:

* Significant alcohol consumption, other causes of liver disease such as viral hepatitis, schistosomiasis, autoimmune, hereditary, drug induced, or decompensated liver cirrhosis.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Group I: included 30 healthy subjects as control. Group II: included 31 patients with NAFLD without liver fibrosis. Group III: included 52 patients with hepatic fibrosis on top of NAFLD.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Serum ferritin in patients with hepatic fibrosis on top of NAFLD | 1 year
  measurement of serum ferritin in patients with hepatic fibrosis on top NAFLD in comparison with normal control and simple steatosis